**Symptom Perception, Behavior, and Outcomes in Older Asthmatics** 

PI: Dr. Juan P Wisnivesky

NCT03646669

Document Date: Jan 18, 2022

## Pilot Test Protocol (Aim 4): Pilot test an intervention to correct under-perception of asthma symptoms in older adults.

Aim 4: Data Analysis: We will compare the baseline characteristics of patients randomized to the intervention vs. control arm using a t-test or chi-square test, as appropriate. Post intervention percent of symptom underperception among groups will be compared using a t-test or Wilcoxon test. In exploratory analyses, we will compare illness (IPQ scores) and medication (BMQ scores) beliefs, adherence (electronic measures, MARS scores), and other SMB (e.g., trigger avoidance) in the PEF intervention vs. control arm. We will also conduct secondary multiple regression analyses adjusting for potential differences in baseline characteristics (including 12-month underperception scores). Power for Aim 4: Based on a sample of 80 participants, the study will have >90% power to identify a clinically meaningful difference of 5 units in symptom perception.